CLINICAL TRIAL: NCT04413591
Title: A Structural HIV Prevention Intervention Targeting High-risk Women
Acronym: EMERALD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00007664; 1R01DA041243 (NIH)
Record Dates: First submitted 2020-05-11; First posted 2020-06-04 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Sex Work
Keywords: Sex work; HIV; STI
MeSH Terms: conditions — Sex Work; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Area (Experimental): Participants are assigned to the intervention area or the control area based on the location they were recruited in.
  Interventions: Behavioral: Community based combination HIV prevention package
- Control Area (No Intervention): Participants are assigned to the intervention area or the control area based on the location they were recruited in.

INTERVENTIONS:
Behavioral: Community based combination HIV prevention package — The intervention compares the efficacy of a community-based comprehensive HIV/STI prevention package compared to standard of care (HIV testing, counseling, and referrals) among Female Sex Workers.
  Arms: Intervention Area

SUMMARY:
The purpose of this study is to assess the effectiveness of a community based combination HIV prevention package, including biomedical, behavioral, and structural services for female sex workers (FSW) in Baltimore, Maryland. This study is a prospective two-group trial comparing the efficacy of a community-based comprehensive HIV/STI prevention package compared to standard of care (HIV testing, counseling, and referrals) among FSWs. Outcomes will be assessed through self-reported illicit drug use and sexual risk behaviors (behavioral) as well as HIV/STI testing (biological).

DETAILED DESCRIPTION:
This study aims:

1. To examine the effect of exposure to community intervention components on HIV/STI risk behaviors (e.g., drug use/unprotected sex), and HIV/STI cumulative incidence over time in FSWs in the intervention (n=275) compared to those in the comparison group (N=175);

   a. to explore the intervention's effects on the risk environment of exotic dance clubs (N=15) over time
2. To examine how socio-structural (e.g., social cohesion, stigma) and structural vulnerability (e.g., financial and housing stability) indicators change and are associated with the biological and behavioral outcomes over time in FSWs in the intervention (n=275) compared to those in the comparison (n=175) group

   a. examine the role of these indicators as mediators of the intervention effect on study outcomes;
3. To examine the intervention's implementation through qualitative (e.g., in-depth interviews) and quantitative (e.g., assessment of program fit, reach, facilitators, barriers, program costs) measures.

3.1 To examine participant knowledge of the COVID-19 crisis as well as the impact of the crisis on their mental, and physical well-being.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older;
* Assigned female at birth and identify with female gender
* Have exchanged sex in Baltimore City at least 3 times in the past 3 months;
* Willing to undergo testing for HIV, gonorrhea, and chlamydia
* Willing to provide locator information.

Exclusion Criteria:

* Inability to provide informed consent in English;
* Women who are determined as too high or drunk;
* Women who are cognitively impaired.
* Currently enrolled in the SAPPHIRE study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned female at birth and identify with female gender
Enrollment: 385 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Change in HIV/STI cumulative incidence over time | Baseline, 6 month, 12 month, 18 month, 24 month visits.
  Participants will be tested for HIV, chlamydia and gonorrhea at each study visit.

SECONDARY OUTCOMES:
Sexual Risk Behaviors | Baseline, 6 month, 12 month, 18 month visits.
  Participants will be asked for detailed information about sexual partners in the last 6 months.
  For each listed partner, the investigators will ask: gender; age; drug use; incarceration history; type of partner (primary, casual, one-time); frequency of sexual activity and condom use; type of sex (oral, vaginal, anal); and if partner had other sexual partners during the time of their sexual involvement. This data collection method allows for calculation of the number of unprotected sexual acts.
Illicit Drug Use | Baseline, 6 month, 12 month, 18 month visits.
  The investigators will ascertain the initiation and frequency of all illicit drugs through the use of a modified NIDA Risk Assessment Battery that has been used and adapted over the past decade.

OTHER OUTCOMES:
Implementation evaluation using SPARC Center client satisfaction surveys | 12-month, 18-month
  SPARC Center client satisfaction surveys will be used to determine the fit, facilitators and barriers, quality, and general experience of women who have used the SPARC Center.
Implementation evaluation using in-depth interviews with SPARC staff and clients | 18 months
  An in-depth interview guide will be developed by experienced study staff and used to interview SPARC guests and staff with the goal of examining program reach, fit, facilitators and barriers, and program costs.
Implementation evaluation using cross-sectional surveys | 18 months
  A cross-sectional survey will be developed by study staff and used to determine the reach of the implementation within the FSW community of southwest Baltimore.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Sherman, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sherman SG, Tomko C, Nestadt DF, Silberzahn BE, Clouse E, Haney K, Allen ST, Galai N. Impact of a Community Empowerment Intervention on Sexually Transmitted Infections Among Female Sex Workers in Baltimore, Maryland. Sex Transm Dis. 2023 Jun 1;50(6):374-380. doi: 10.1097/OLQ.0000000000001781. Epub 2023 Feb 8. PMID 36749851
- [Derived] Silberzahn BE, Tomko CA, Clouse E, Haney K, Allen ST, Galai N, Footer KHA, Sherman SG. The EMERALD (Enabling Mobilization, Empowerment, Risk Reduction, and Lasting Dignity) Study: Protocol for the Design, Implementation, and Evaluation of a Community-Based Combination HIV Prevention Intervention for Female Sex Workers in Baltimore, Maryland. JMIR Res Protoc. 2021 Apr 16;10(4):e23412. doi: 10.2196/23412. PMID 33861210